CLINICAL TRIAL: NCT07093905
Title: Prospective, Randomized Study Comparing General Anesthesia Combined With Locoregional Anesthesia to Locoregional Anesthesia Alone for Arthroscopic Rotator Cuff Repair.
Brief Title: Study Comparing Two Anesthetics for Arthroscopic Rotator Cuff Repair
Acronym: ALRAGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00971-48
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, randomized, open-label, multicenter study comparing two analgesic strategies
Masking Description: open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locoregional anesthesia (Experimental): patients will benefit from locoregional anesthesia alone by means of an interscalene block of the brachial plexus.
  Interventions: Procedure: arthroscopy of the shoulder rotator cuff
- Locoregional anesthesia + general anesthesia (Active Comparator): patients will benefit from general anesthesia as well as locoregional anesthesia via an interscalene block of the brachial plexus.
  Interventions: Procedure: arthroscopy of the shoulder rotator cuff

INTERVENTIONS:
Procedure: arthroscopy of the shoulder rotator cuff — minimally invasive surgical procedure in which a camera (arthroscope) is inserted into the shoulder joint

SUMMARY:
The purpose of this study is to to compare the post-anesthetic recovery time to awake consciousness and hemodynamic and ventilatory capacities for discharge from the Post-Interventional Monitoring Room in patients admitted for shoulder rotator cuff arthroscopy (using local anesthesia versus general anesthesia + local anesthesia).

DETAILED DESCRIPTION:
This is a prospective, comparative, randomized, open-label, multicenter study comparing two analgesic strategies used in outpatient, routine surgery.

The study population is composed of adult patients with complete or partial rotator cuff tears requiring reconstructive surgery under anesthesia at Hôpital Privé Clairval or Clinique Monticelli-Vélodrome.

Patients will be seen three times: at inclusion (during the preoperative consultation with the anesthetist), on the day of surgery (hospitalization), and at the follow-up visit (during the postoperative consultation with the surgeon). They will also be contacted by telephone on D1, D3 and D15 to optimize their follow-up. The duration of each patient's participation is approximately one month.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with surgically repairable complete or partial rotator cuff tears;
* American Society of Anesthesiologists Class I to III;
* Patient able to understand study information;
* Patient willing to accept study evaluations and follow-up visits;
* Affiliation with a social insurance plan;
* Patient having been informed and having agreed to participate in the study by signing an informed consent form.

Exclusion Criteria:

* Contraindication to general or locoregional anesthesia;
* Chronic opioid use;
* Patient unable to understand study information (linguistic, psychological, cognitive, etc.);
* Patient unable to answer a self-questionnaire;
* Patient participating in or being excluded from another interventional research study;
* Pregnant or breast-feeding women;
* Protected patient (under legal protection, guardianship or deprived of liberty by judicial or administrative decision).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
length of stay in the Post-Interventional Monitoring Room | Day 0
  The primary endpoint is the length of stay in the Post-Interventional Monitoring Room from discharge from the operating room to an Aldrete score > 8 leading to discharge from the Post-Interventional Monitoring Room.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Clairval, Marseille, France